CLINICAL TRIAL: NCT01357954
Title: The Efficacy of Targeted Training on the Postural Control and Gross Motor Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Derek Curtis, Research Physiotherapist, Hvidovre University Hospital., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVH-DJC-1-2011
Record Dates: First submitted 2011-05-06; First posted 2011-05-23 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy
Keywords: Postural control; Targeted Training; Gross motor function; Cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Training (Experimental)
  Interventions: Other: Targeted Training
- Control (Other)
  Interventions: Other: Regular physiotherapy

INTERVENTIONS:
Other: Regular physiotherapy — The child's regular physiotherapy
  Other Names: Physiotherapy
  Arms: Control
Other: Targeted Training — Targeted training, 5 days a week for 6 months, up to 30 minutes a day
  Other Names: The Movement Centre
  Arms: Targeted Training

SUMMARY:
The project aims to test the effectiveness and explore the possibility of performing a novel therapeutic approach, targeting to increase strength and coordination around the trunk, giving a more active and functional seating and head control in those children with cerebral palsy (CP) who are wheelchair users. The project will also try to determine the muscle physiological effect of treatment using indirect measures of strength in the spinal musculature.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CP made by a neuro-pediatric physician experienced in assessment and diagnosis of CP
* GMFCS level III, IV and V,
* the child cannot walk without assistance,
* age 2-15 year,
* no joint deformity or contracture around the "Targeted" joint
* not a candidate for surgery or other medical treatment that affects motor skills while participating in the project
* trunk control problems.

Exclusion Criteria:

* uncontrolled epilepsy
* surgery within 12 months of the study start
* Botulinum toxin within 2 months of study start
* Lack of personnel resources to treat the child at their school/kindergarten

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Gross Motor Function Measure at 6 months | Baseline, 6 months

SECONDARY OUTCOMES:
Change from baseline in Pediatric Evaluation of Disability Inventory (PEDI)at 6 months | Baseline, 6 months
Change from baseline in thickness of the erector spinae muscles measured with ultrasound at 6 months | Baseline, 6 months
Change from baseline in seated sway at 6 months | Baseline, 6 months
Degree of achievement of a goal set at baseline using a modified Goal Attainment Scale (GAS) | 6 months
Change from baseline in Pediatric Evaluation of Disability Inventory (PEDI)at 12 months | Baseline, 12 months
Change from baseline in thickness of the erector spinae muscles measured with ultrasound at 12 months | Baseline, 12 months
Change from baseline in seated sway at 12 months | Baseline, 12 months
Degree of achievement of a goal set at baseline using a modified Goal Attainment Scale (GAS) | 12 months
Change from baseline in Gross Motor Function Measure at 12 months | Baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Curtis, PT MSc, Principal Investigator — Hvidovre University Hospital; Stig Sonne-Holm, Dr Med, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark